CLINICAL TRIAL: NCT00744458
Title: A Prospective Randomised Trial Comparing Three Interventions to Improve Treatment Adherence Among Patients With Arterial Hypertension or Diabetes in Rural Cameroon (TAHADIRA-trial 1)
Brief Title: Treat Arterial Hypertension and Diabetes in Rural Africa
Acronym: TAHADIRA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cooperation Afrique (Other)
Responsible Party: Niklaus Labhardt, Cooperation Afrique
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: TAHADIRA
Record Dates: First submitted 2008-08-29; First posted 2008-09-01 (Estimated); Last update posted 2010-05-27 (Estimated); Status verified 2009-08

CONDITIONS: Diabetes; Arterial Hypertension
Keywords: Primary Health care in rural Africa; Chronic non-communicable diseases; Patient Compliance; Treatment adherence
MeSH Terms: conditions — Diabetes Mellitus; Hypertension; Noncommunicable Diseases; Patient Compliance; Treatment Adherence and Compliance

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Active Comparator)
  Interventions: Other: Treatment contract
- 2 (Active Comparator)
  Interventions: Other: Treatment contract; Other: Tracing and recall at home by a community worker
- 3 (Active Comparator)
  Interventions: Other: Treatment contract; Other: Incentive

INTERVENTIONS:
Other: Treatment contract — Patients signs in for a agreement - to respect a regular follow-up at the health facility.
Other: Tracing and recall at home by a community worker — The local health committee sends out a member to trace the patient and to motivate him to take up again regular treatment visits.
  Arms: 2
Other: Incentive — Incentive by giving free treatment after a 4-month regular follow-up
  Arms: 3

SUMMARY:
The purpose of this study is to determine the efficacy of three different interventions to improve treatment adherence among patients with arterial hypertension or diabetes in rural Cameroon.

DETAILED DESCRIPTION:
Non communicable chronic diseases such as arterial hypertension (AH) and diabetes (DM) are a great burden for public health in Cameroon. However, outside the main cities access to appropriate diagnosis and treatment of these health-conditions is still very poor.

The Swiss NGO "Fondation Coopération Afrique" started in 2007 a program to integrate chronic disease management with focus on AH and DM into the primary health care system of peripheral non-physician health facilities in a rural area of Central Cameroon. A first evaluation after one year revealed very low treatment adherence among the newly diagnosed patients as the main challenge.

In order to improve patient's adherence we expose them randomly to one of three interventions:

The first intervention consists in a written agreement on long-lasting therapy (treatment contract). Patients get information about the importance of a regular long term treatment and personal engagement to follow treatment and clinical controls regularly.

The second intervention introduces in addition to the treatment contract a reminder system. In case of follow-up failure a community worker traces the patient to recall the visit at the health centre.

The third intervention consists of the treatment contract combined with a financial incentive in form of one month free treatment after four months of regular follow-up.

We allocated randomly one of the three interventions to each health center.

ELIGIBILITY:
Inclusion Criteria:

* Patients with newly diagnosed arterial hypertension or non insulin dependent diabetes type 2 which require treatment and can be treated in the health centre
* Informed consent by the patient

Exclusion Criteria:

* Patient already under treatment
* Patients who need to be referred to a hospital
* No informed consent by the patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 223 (Actual)
Dates: Start 2008-08; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with regular follow-up one year after the treatment was started | One patient year

SECONDARY OUTCOMES:
Percentage of missed control-visits | One patient year
Treatment response of diabetic patients (fasting blood glucose) | One patient year
Treatment response of patients with arterial hypertension (blood pressure) | One patient year

CONTACTS AND LOCATIONS:
Overall Officials: Engelbert Manga, MD, MPH, Study Director — Medical district officer of Mfou, Ministry of public health of Cameroon; Niklaus D Labhardt, MD, Principal Investigator — Representant of the foundation Coopération Afrique, Switzerland; Beat Stoll, MD, MPH, Study Chair — Institute of social and preventive medicine, University of Geneva, Switzerland
Locations (1):
- Medical districts of Mfou, Mbankomo Obala and Esse in Central Cameroon, Divisions of Mefou and Lékié, Central Province, Cameroon